CLINICAL TRIAL: NCT04249544
Title: Cognitive and Neural Mechanisms of Impaired Social Decision-Making in Parkinson's Patients Taking Dopamine Agonists
Brief Title: Social Decision Making in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Darby, Assistant Professor of Neurology, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Social Decision Making in PD; W81XWH-19-1-0782 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Impulsive behavior; Social decision making; Moral decision making; dopamine agonists
MeSH Terms: conditions — Parkinson Disease; Impulsive Behavior | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Impulsive group, placebo then pramipexole (Experimental): half of the impulsive group will first get the placebo on the first day and pramipexole on the second day
  Interventions: Drug: Pramipexole; Drug: Placebo
- Impulsive group, pramipexole then placebo (Experimental): half of the impulsive group will first get the pramipexole on the first day and the placebo on the second day
  Interventions: Drug: Pramipexole; Drug: Placebo
- Non-impulsive group, placebo then pramipexole (Experimental): half of the non-impulsive group will first get the placebo on the first day and the pramipexole on the second day
  Interventions: Drug: Pramipexole; Drug: Placebo
- Non-impulsive, pramipexole then placebo (Experimental): half of the non-impulsive group will first get the pramipexole on the first day and the placebo on the second day
  Interventions: Drug: Pramipexole; Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole — 1mg of pramipexole
Drug: Placebo — 1mg equivalent of placebo

SUMMARY:
Impulsive and compulsive behaviors occur in up to 46% of Parkinson's Disease (PD) patients taking dopamine agonist (DAA) medications. While these abnormal social behaviors have been studied in other neurodegenerative disorders, the true incidence of social problems, and the relationship to dopamine therapy, in PD patients remains unknown. This study is aiming to determine if dopamine agonists alter social decision-making and to determine if impaired social decision-making relates to dopamine-induced mesolimbic network dysfunction in PD patients. The protocol will include a screening visit, and on-DAA visit, and an off-DAA visit. For both the on and off DAA visits, participants will continue taking Carbidopa-Levodopa, but will withdrawal off of other PD related medications. Both visits will include an MRI, fMRI shock task, questionnaires to be filled out by other the participant and the caregiver, moral-decision making computer tasks, and the Unified Parkinsons Disease Rating Scale (UPDRS) part II and III. For the on-DAA visit, participants will take Pramipexole. For the off-DAA visit, participants will receive a placebo. Participants will remind blinded to which medication they are receiving that day and will be counterbalanced such that all participants will not take the Pramipexole or placebo on the same days.

DETAILED DESCRIPTION:
Impulsive and compulsive behaviors occur in up to 46% of Parkinson's Disease (PD) patients taking dopamine agonist (DAA) medications. While these abnormal social behaviors have been studied in other neurodegenerative disorders, the true incidence of social problems, and the relationship to dopamine therapy, in PD patients remains unknown. This study is aiming to determine if dopamine agonists alter social decision-making and to determine if impaired social decision-making relates to dopamine-induced mesolimbic network dysfunction in PD patients. The protocol will include a screening visit, and on-DAA visit, and an off-DAA visit. For both the on and off DAA visits, participants will continue taking Carbidopa-Levodopa, but will withdrawal off of other PD related medications to reduce circulating drugs and residual drug effects. Both visits will include an MRI, fMRI shock task, questionnaires to be filled out by other the participant and the caregiver, moral-decision making computer tasks, and the Unified Parkinson's Disease Rating Scale (UPDRS) part II and III. For the on-DAA visit, participants will take Carbidopa-Levodopa 1 hour before the scan and will take 1mg of Pramipexole 1 hour before the scan. For the off-DAA visit, participants will take Carbidopa-Levodopa 1 hour before the scan and will take a placebo 1 hour before the scan. Participants will remind blinded to which medication they are receiving that day and will be counterbalanced such that all participants will not take the Pramipexole or placebo on the same days.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-80
* Ability to give informed consent
* Idiopathic Parkinson's disease
* Currently taking dopamine agonist therapy
* Mild symptom severity (Hoehn & Yahr ≤ 3)
* Disease duration of <12 years
* Demonstrated positive response to dopamine therapy

Exclusion Criteria:

* Medications classes that influence GABA concentrations: benzodiazepines, cholinesterase inhibitors, antipsychotics, opioids, and MAO inhibitors
* History of substance abuse or use of any psychostimulants (other than caffeine) in the last 6 months or more than 4 times in lifetime
* Current tobacco (or nicotine use) or alcohol intake greater than 8 ounces of whiskey or equivalent per week
* Comorbid neurological disorders (e.g., stroke, peripheral neuropathy, seizure disorder) or history of head trauma (other than a single concussion)
* Unstable medical condition, [e.g., diabetes or pulmonary disease, significant medical condition, including high blood pressure (systolic B.P. > 135, Diastolic B.P. > 85), or any hepatic, renal, cardiovascular, hematological, endocrine or ophthalmological condition]
* History of major psychiatric illness (including any affective disorder, substance use disorder, psychotic disorder, or eating disorder)
* Dementia
* Deep brain stimulation
* Contraindications to 3 Tesla MRI, e.g., extreme obesity, claustrophobia, cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, tattoos with iron pigment and metallic body inclusions or other metal implanted in the body
* Dyskinesia or tremor that would cause severe motion artifact during MRI scan
* Clear indication of secondary gain

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The change in a harm aversion cognitive moral decision-making task | two weeks
  change in harm aversion from off drug visit to on drug visit
change in blood flow in the ventral striatum per ASL images | two weeks
  change in CBF from off drug visit to on drug visit

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Darby, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT04249544/ICF_000.pdf